CLINICAL TRIAL: NCT00042601
Title: A Single Center, Randomized, Double-blind, Placebo-controlled, Two-period, Crossover Study Evaluating the Acute Effect of Pramlintide on Satiety and Food Intake in Normal-weight and Obese Non-diabetic Subjects and in Insulin Treated Subjects With Type 1 and Type 2 Diabetes Mellitus
Brief Title: Evaluation of the Effect of Pramlintide on Satiety and Food Intake
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 137-149
Record Dates: First submitted 2002-08-01; First posted 2002-08-05 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — pramlintide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): A clear, colorless, sterile solution for SC injection manufactured by Amylin Pharmaceuticals, Inc. Placebo solution is the same, sterile preserved formulation, except the active ingredient, pramlintide, is omitted.
  Interventions: Drug: Placebo
- Pramlintide (Active Comparator): Pramlintide acetate (AC137) injection is a clear, colorless, sterile solution for SC injection manufactured by Amylin Pharmaceuticals, Inc. It consists of pramlintide (AC137) 0.6 mg/mL in sodium acetate buffer, pH 4.0, containing 43 mg/mL mannitol as an iso-osmolality modifier and 2.25 mg/mL metacresol as a preservative.
  Interventions: Drug: Pramlintide acetate

INTERVENTIONS:
Drug: Pramlintide acetate — Pramlintide injection will be supplied in 5-mL multidose glass vials with rubber stoppers.
  Arms: Pramlintide
Drug: Placebo — placebo injection will be supplied in 5-mL multidose glass vials with a rubber stopper
  Arms: Placebo

SUMMARY:
This is a single center, randomized, blinded, placebo-controlled, two-period, cross-over study to evaluate the effect of pramlintide on satiety and food intake in normal-weight and obese non-diabetic subjects and in insulin-treated subjects with type 1 and type 2 diabetes.

ELIGIBILITY:
For Healthy Volunteers:

•BMI >=20 to <=25kg/m2 or >=30 to <=40 kg/m2

For Subjects with Type 1 or Type 2 Diabetes:

* Treated with insulin for at least 6 months prior to screening
* HbA1c value between 6.5-10% inclusive
* BMI between 20-40kg/m2

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2002-07; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Change in satiety of participants on Pramlintide | 2 Weeks
  To assess the acute effect of pramlintide administered subcutaneously (SC) on satiety in normal-weight and obese non-diabetic subjects and in insulin-treated subjects with type 1 and type 2 diabetes. To be measured by Total caloric intake, macronutrient intake (carbohydrate, fat, protein, and other), duration of buffet meal, aand satiety data measured via a satiety assessment at Period 1 (Visit 2) and Period 2 (Visit 3).
Change in food intake of participants on Pramlintide | 2 Weeks
  To assess the acute effect of pramlintide administered SC on food intake in normal-weight and obese non-diabetic subjects and in insulin-treated subjects with type 1 and type 2 diabetes. To be measured by Total caloric intake, macronutrient intake (carbohydrate, fat, protein, and other), duration of buffet meal, aand satiety data measured via a satiety assessment at Period 1 (Visit 2) and Period 2 (Visit 3).

SECONDARY OUTCOMES:
Effect of pramlintide on postprandial metabolic and hormonal responses | 2 Weeks
  To assess the acute effect of pramlintide administered SC on postprandial metabolic and hormonal responses [glucose, triglycerides, total cholesterol, insulin, cholecystokinin (CCK), and glucagon-like peptide (GLP-1)] in normal-weight and obese non-diabetic subjects and in insulin-treated subjects with type 1 and type 2 diabetes. To be measured by the calculation of both absolute and incremental plasma analyte concentration profiles.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Adelaide Hospital, Adelaide, South Australia, Australia